CLINICAL TRIAL: NCT05722756
Title: Comparison of Rehabilitation Techniques: Vojta vs Vojta and Craniosacral Therapy, in Children With Central Nervous Coordination Disorders.
Brief Title: The Effect of Craniosacral Therapy as Additive Procedure.
Acronym: COREHNERV
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 108/2019
Record Dates: First submitted 2023-01-20; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Central Nervous System Diseases
Keywords: children; rehabilitation; central nervous system; Vojta therapy; cranio-sacral therapy; reflex locomotion
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: treated with Vojta therapy
- group B: treated with Vojta therapy combined with craniosacral therapy
  Interventions: Other: craniosacral therapy

INTERVENTIONS:
Other: craniosacral therapy — subtle form of applied touch, type of osteopathy
  Groups: group B

SUMMARY:
This observational, retrospective study has shown, that the addition of craniosacral therapy to the Vojta method has improved the effects of the therapy in 6 months follow-up period. The chance for improvement was 9.42 times higher in Vojta + craniosacral group compared to the group conducted only with Vojta method.

The study results suggest that the craniosacral procedure should be considered as an additive regimen to the Vojta method in the therapy of children with central coordination disorders (CCD) . More data is still needed to improve the rehabilitation process in this group of patients.

DETAILED DESCRIPTION:
The aim of the retrospective, observational study was the comparison between the effectiveness of Vojta therapy used alone and its combination with craniosacral therapy after 6 months of the therapy.

Data for analysis was from one Rehabilitation Center and covered the observation period: January 1, 2014 - November 30, 2019. The data was analyzed for the purpose of the study between January 1, 2022 - July 1, 2022.

To assess the effectiveness of the mentioned rehabilitation models for the children with central coordination disorders (CCD), the neurological status of the patient, expressed as the number of abnormal reactions (Vojta tests), at the beginning (W0) and after 6 months (W6) of the therapy was recorded blindly, based on the individual's records (collected previously for the purpose of the other study). Children who had completed six months of therapy and had efficacy results documented in their medical records were divided into group A (children treated with Vojta therapy alone) and group B (children treated with Vojta therapy combined with craniosacral therapy). Information about: the age at which the children started therapy, the APGAR score at the first minute of their life, the week in which they were born, mode of delivery, sex, birth weight, mother's age at delivery and duration of breastfeeding, was also collected to compare the groups.

Finally data from 32 children in group A and 19 children in group B was analyzed.

ELIGIBILITY:
Inclusion criteria:

* CCD (central coordination disorders) diagnosis based on the paediatrician's opinion with a decision that the child needs rehabilitation;
* a score of 8- 10 on the APGAR scale in the first minute of life;
* no major birth defects documented that can push the diagnosis into the diagnosis of genetic disorders;
* the age of the child at the time of the assessment of its eligibility for rehabilitation: 1-6 months (of life), calculated based on completed months of life;
* available information regarding an abnormal result of the Vojta test, defined as at least 6 abnormal reactions (marked as abnormal [AN], or delayed [OP] in the test report) with abnormal muscle tension, which indicates moderate to severe CCD;
* available information regarding the first medical examination (during the first visit (W0)), and a follow-up visit after 6 months (W6) on the determined date, maintaining the defined timeframe (5.5-6 months after W0).

Exclusion criteria (medical history was excluded from the analysis even if one of the following exclusion criteria was met):

* children who obtained a score of < 8 points on the APGAR scale in the first minute of life;
* suspicion of any major (significant) birth defect, congenital defect syndrome (e.g. Down syndrome, Sotos syndrome) and/or indications for consultation at Genetics Clinic based on paediatric records;
* age < 1 month or > 6 months;
* < 6 abnormal reactions during the Vojta test at the first eligibility visit, which indicates mild or very mild CCD.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with confirmed CCD (central coordination disorders), between 1-6 months of age
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in the number of abnormal reactions (assessed by the Vojta tests) | 6 months
  improvement: fewer number of the abnormal reactions present when compare to the first visit no improvement- at least the same number (or more) of abnormal reactions present when compare to the first visit

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: after publication, no limit
Access Criteria: to everyone via the link below
URL: https://ppm.umed.wroc.pl/info/researchdata/UMW4043bfe107e64b6a83a72d78286d80f1/